CLINICAL TRIAL: NCT06777277
Title: Cognitive-Behavioural Couple Therapy for Sexual Interest/Arousal Disorder
Acronym: CBCT for SIAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dalhousie University (Other)
Collaborators: Université de Montréal (Other); University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-7379; 496676 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2025-01-06; First posted 2025-01-15 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-11

CONDITIONS: Sexual Interest/Arousal Disorder
Keywords: cognitive-behavioral couple therapy; Emotion regulation; Sexual dysfunction; Female sexual interest/arousal disorder; DSM-5
MeSH Terms: conditions — Emotional Regulation; Sexual Dysfunction, Physiological | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: The randomized clinical trial will evaluate the efficacy of a novel 16-session online CBCT for an inclusive sample of women with SIAD compared to a waitlist control group. Couples in the waitlist control group will complete all questionnaires at the equivalent timepoints as the experimental group. At the end of the 6-month follow-up, waitlist couples will be offered CBCT free-of-charge.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will be randomized to one of the two study arms before treatment initiation (max 2 weeks delay) using a stratified method, based on the treatment site. Assignments will be made by a free randomization software (www.studyrandomizer.com). In each site, allocation will be computer-generated randomly using permuted blocks of size 6 (fixed) to maintain equilibrium between the two conditions (treatment and control). This procedure ensures that the personnel conducting evaluations will not be aware of participant condition and that the PIs will not influence the randomization process. Data analysts will be masked until the end of all analyses. Participants will be instructed not to reveal the condition they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBCT for SIAD (Experimental): 16 sessions of cognitive-behavioural couple therapy.
  Interventions: Other: Cognitive-behavioral therapy
- Waitlist (No Intervention): Description: The investigators selected a waitlist control comparison as the first step to establishing efficacy of the CBCT because there are no existing empirically validated couple-based treatments available for SIAD.

INTERVENTIONS:
Other: Cognitive-behavioral therapy — The intervention will be delivered in 16, 60-minute sessions (1st session 90 mins). The treatment manual was informed by a 12-session (75 min each) CBCT developed by our team for genito-pelvic pain. The SIAD manual focuses on empirically supported interpersonal factors relevant to SIAD, informed by the Interpersonal Emotion Regulation Model of women's sexual dysfunction. The goals of the CBCT are to: (1) re-conceptualize low sexual desire/arousal as multidimensional in which both partners affect and are affected by the SIAD symptoms (2) modify and/or accept those factors that are associated with low sexual desire/arousal to increase adaptive coping, facilitate sexual desire/arousal, and reduce sexual distress, (3) as per our theoretical model, improve couple interactions related to sexuality (e.g., communication, intimacy) via enhanced emotion regulation, and (4) consolidate skills.
  Arms: CBCT for SIAD

SUMMARY:
Sexual health is a fundamental aspect of quality of life; a satisfying sexual relationship is linked to better physical, psychological, and relationship health and well-being. In fact, people who maintain a satisfying, active sex life over time live longer than those who report lower sexual frequency and satisfaction. Yet problems with sexual function are extremely common, especially for women: chronic difficulties with sexual desire and/or arousal that are personally upsetting-Sexual Interest/Arousal Disorder (SIAD)-affects 7% to 23% of the general population. SIAD is linked to more healthcare costs, depressive symptoms and anxiety, and lower relationship satisfaction. Experts suggest that relationship factors play a critical role in SIAD and couple-based sex therapy is a common approach used by clinicians. However, there are no treatment options available for couples that have been tested in research to confirm that they work. The goal of this three-centre randomized clinical trial is to evaluate the efficacy of a novel 16-session cognitive-behavioural couple therapy (CBCT), offered online to increase accessibility, for an inclusive sample of women with SIAD compared to a waitlist control group. The investigators expect that, compared to a waitlist control group, CBCT will lead to greater improvements in SIAD symptoms (e.g., higher sexual desire/arousal, lower sexual distress) and better sexual, relational, and psychological adjustment for both partners at post-treatment and 6-months later. Given that less than a third of those affected by SIAD access treatment, this study addresses the urgent need for an accessible couple-based treatment for the most common sexual dysfunction. Results will be used by clinicians to provide couples with a scientifically based, accessible treatment option, that will improve their sexual, relationship, and psychological health.

DETAILED DESCRIPTION:
Background and Importance. Sexual health is a fundamental aspect of overall quality of life; a satisfying sexual relationship is associated with better physical, psychological, and relationship health and well-being. In fact, people who maintain a satisfying, active sex life over time live longer than those who report lower sexual frequency and satisfaction. Yet problems with sexual function are extremely common, especially for women: persistent difficulties with sexual desire and/or arousal that are personally distressing-Sexual Interest/Arousal Disorder (SIAD9)-affects 7% to 23% of the general population. SIAD is linked to greater healthcare costs, depressive symptoms, and lower relationship satisfaction. Sexual desire-the key component in SIAD-is thought to be embedded in, and influenced by, interpersonal factors, more so for women than for men. Although theoretical and clinical models suggest a significant role for interpersonal processes in SIAD, there is a striking neglect of these factors in available treatments. Couple-based sex therapy is commonly used by clinicians, but no study to date has assessed its efficacy for SIAD. The current proposal builds on our ongoing CIHR-funded work examining interpersonal factors in SIAD, as well as the results of our pilot study.

Aims. The primary aim of this three-centre randomized clinical trial is to test the prediction that a novel cognitive-behavioural couple therapy (CBCT) delivered online will yield significantly greater improvements in primary outcomes of sexual desire and sexual distress for women and individuals with SIAD post-treatment and 6-months later, compared to a waitlist control group. Our secondary aim is to test the prediction that couples receiving CBCT will report greater improvements in sexuality, relationship, and psychological outcomes relative to the control group.

Methods/Approach/Expertise. The investigators will: (1) recruit an inclusive sample of 170 women diagnosed with SIAD via a clinical interview, and their partners; (2) randomize couples to either the 16-session CBCT or a waitlist control group; (3) have couples complete standardized, self-report measures at pre-treatment, post-treatment, and 6-month follow-up as well as approximately every 4 weeks during the treatment period; (4) test the efficacy of CBCT compared to the control group. Procedures will take place at Dalhousie University, Université de Montréal, and the University of British Columbia.

Expected Outcomes. This clinical trial addresses the urgent need for an empirically validated, accessible, couple-based treatment for the most prevalent sexual dysfunction-SIAD. Results will be used by clinicians to provide affected couples with a scientifically-based treatment option that will improve their sexual, relationship and psychological well-being.

ELIGIBILITY:
Inclusion Criteria:

* One member of the couple must identify as a cisgender woman, a trans woman, or a gender diverse person assigned female at birth;
* One member of the couple must meet diagnostic criteria for SIAD;
* Both partners must be fluent in English or French;
* Both partners must be in a committed, cohabiting relationship for at least one year (with a partner of any gender/sex).

Exclusion Criteria:

* Pregnancy, breastfeeding or one year postpartum;
* No prior sexual experience;
* Severe relational distress or conflict as determined by baseline measures and interview;
* Are currently undergoing treatment for SIAD, or are in couple or sex therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Since this study is about women's low sexual desire and/or arousal, the investigators are recruiting couples in which one member is a cisgender woman, trans woman, or gender diverse person assigned female at birth.
Enrollment: 170 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Sexual Desire | A. At baseline (after enrolment in the study) B. During treatment (approximately 4, 8, 12 and 16 weeks after baseline) C. At post-treatment (approximately 18 weeks after baseline) D. At 6-month follow-up (6M after post-treatment)
  As a core symptom of SIAD, partner-focused dyadic sexual desire will be assessed using the 7-item subscale of the Sexual Desire Inventory. This subscale measures interest in sexual activity, including one's thoughts on approaching or being responsive to sexual stimuli with a partner, in a Likert-type response format (e.g., 1 = not at all, 7 = a lot). Higher scores indicate greater partner-focused dyadic sexual desire. For the in-treatment surveys, a shorter version of the Sexual Desire Inventory-2, including two items, will be used to minimize participant burden. This version has been used in prior studies and showed adequate psychometric properties.
Sexual Distress | A. At baseline (after enrolment in the study) B. During treatment (approximately 4, 8, 12 and 16 weeks after baseline) C. At post-treatment (approximately 18 weeks after baseline) D. At 6-month follow-up (6M after post-treatment)
  As a core symptom of SIAD, sexual distress will be measured with the 5-item Sexual Distress Scale-SF (SDS-SF). Using a 5-point Likert scale, participants rate how frequently (e.g., 1 = never, to 5 = always) they experience an emotion or sexuality related problem. These items showed greatest function at the item level, greatest contribution to the scale's reliability, and good capacity to discriminate between participants with distressing sexual problems and those without distressing sexual problems. This measure is valid regardless of whether participants are sexually active. For the in-treatment surveys, the three-item version of the SDS-SF will be used to minimize participant burden. It has been used in previous studies and showed adequate psychometric properties.

SECONDARY OUTCOMES:
Sexual Satisfaction | A. At baseline (after enrolment in the study) B. During treatment (approximately 4, 8, 12 and 16 weeks after baseline) C. At post-treatment (approximately 18 weeks after baseline) D. At 6-month follow-up (6M after post-treatment)
  The Global Measure of Sexual Satisfaction (GMSEX) assesses overall sexual satisfaction. This scale consists of five items assessing a subjective evaluation of the sexual relationship on five 7-point dimensions: good vs. bad, pleasant vs. unpleasant, positive vs. negative, satisfying vs. unsatisfying, and valuable vs. worthless. Ratings are summed such that possible scores range from 5 to 35, with higher scores indicating greater sexual satisfaction. For the in-treatment surveys, a one-item measure of sexual satisfaction will be used to minimize participant burden. Previously used by our team and showing adequate psychometric properties, the single-item measure asks participants to rate, on a scale of 1 (Very dissatisfied) to 5 (Very satisfied), their answer to the following question: "Since the last survey, how satisfied have you been with your relationship with your partner?".
Relationship Satisfaction | A. At baseline (after enrolment in the study) B. At post-treatment (approximately 18 weeks after baseline) C. At 6-month follow-up (6M after post-treatment)
  It will be assessed with the 16-item Couples Satisfaction Index. Participants will rate their relationship on a number of factors. For example, participants will indicate how happy they are with their relationship, how frequently they disagree with their partner, and how they feel their relationship compares to others. For the in-treatment surveys, participants will fill the four-item shorter version.
Relationship intimacy | A. At baseline (after enrolment in the study) B. At post-treatment (approximately 18 weeks after baseline) C. At 6-month follow-up (6M after post-treatment)
  Intimacy will be measured using 9 items on a 7-point scale (1 = not at all, 7 = a lot) where participants rate in general how much they perceived their partner to be responsive, self- and partner-disclosure of private thoughts and feelings and the level of overall intimacy they feel in their relationship.
Psychological adjustment | A. At baseline (after enrolment in the study) B. At post-treatment (approximately 18 weeks after baseline) C. At 6-month follow-up (6M after post-treatment)
  It will be measured using the Hospital Anxiety and Depression Scale. This 14-item measure includes two subscales: depression (seven items) and anxiety (seven items). Using a time reference of the last 7 days, participants score each item on a scale from 0 (e.g., Not at all) to 3 (e.g., Most of the time), with higher scores indicating greater severity of symptoms. This measure has been shown to have good reliability and validity.
Post-treatment satisfaction and participant global ratings of improvement | A. At post-treatment (approximately 18 weeks after baseline) B. At 6-month follow-up (6M after post-treatment)
  Post-treatment satisfaction will be measured using 3 items asking participants to (a) rate on a scale from 0 to 10 their global satisfaction towards the treatment received, (b) whether there is anything else they would like to share about their experience in this treatment, (c) their satisfaction with completing couple therapy via virtual care (on Zoom) on a scale from 0 to 10.
  Global ratings of improvement will be measured using 3 items assessing on a scale of 0 (deterioration) to 5 (complete recovery) (a) if there has been an improvement in their sexual desire and/or arousal difficulties following the treatment, (b) if there has been an improvement in distress (negative emotions) about their sex life following the treatment, (c) if there has been an improvement in the overall quality of their sex life following the treatment.

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - University of British Columbia, Vancouver, British Columbia
  - Dalhousie University, Halifax, Nova Scotia
  - Université de Montréal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No